CLINICAL TRIAL: NCT04782570
Title: Nicht-invasive Hirnstimulation in Der Psychotherapie Von Angsterkrankungen
Brief Title: Psychotherapy of Anxiety Disorders With Noninvasive Brain Stimulation - Using Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wuerzburg45/20-am; PAN_VR (Other: Clinic for Psychiatry)
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Phobia
Keywords: VR; Exposure therapy; Acrophobia; rTMS; PFC
MeSH Terms: conditions — Phobic Disorders; Acrophobia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum TMS (Experimental): ITBS (intermittent Theta Burst Stimulation) over left frontal cortex
  Interventions: Device: Verum TMS
- Sham TMS (Sham Comparator): Sham TMS over left frontal cortex
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Verum TMS — Intensity of 100% of the resting motor threshold with iTBS. 600 stimuli applied in bursts of three pulses at 50 Hz given every 200 ms. iTBS will be applied 20 times for 2 s every 10 s.
  Other Names: Cool-B70 A/P, MagPro X100, MagVenture®, Denmark
  Arms: Verum TMS
Device: Sham TMS — Sham stimulation with same protocol, but without magnetic stimulation
  Other Names: Cool-B70 A/P, MagPro X100,, MagVenture®, Denmark
  Arms: Sham TMS

SUMMARY:
The aim of the study is to transfer the rTMS stimulation protocol by Raij et al. (2018) into a therapeutic setting to improve exposure therapy in acrophobic patients. The quasi-randomized, placebo-controlled and double-blinded study will include 88 patients with height phobia (according to DSM 5). All participants will perform two exposure sessions in virtual reality (VR). Before exposure therapy, one group will receive verum rTMS of the left frontal cortex, which is indirectly functionally linked to the ventromedial prefrontal cortex (Raij et al., 2018). The control group will receive sham stimulation. A structural MRI and a TMS navigation system will be used for precise localization of the left FC. Anxiety symptoms will be measured using subjective ratings (e.g. Acrophobia Questionnaire) and the behavioural approach task (BAT) in VR and in real life before and after the treatment, and at 6 months follow-up. Furthermore, blood samples will be collected before rTMS and after exposure treatment to assess epigenetic and gene expression based changes.

DETAILED DESCRIPTION:
The following hypotheses are derived:

1. Patients with acrophobia, who receive an active rTMS of the left FC before VRET, show a significantly stronger reduction of phobic symptoms immediately after exposure therapy, compared to the sham stimulation group.
2. Patients with acrophobia, who receive an active rTMS of the left FC before VRET, show a significantly greater increase in approach behavior and significantly less distress during the BAT immediately after exposure therapy, compared to the sham stimulation group.
3. The postulated differences in hypotheses 1 and 2 are still detectable at follow-up after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Acrophobia (according to DSM-5)
* Right handed
* German native speaker
* Written informed consent

Exclusion Criteria:

* Neurological and/or severe physical illnesses
* Comorbid Axis I disorder (other than phobias)
* Pretreated phobia of heights
* Use of tricyclic antidepressants, antipsychotics, or other substances that increase cerebral seizure susceptibility
* Craniocerebral injuries, head surgery
* Epileptic seizures, or family history of epilepsy
* Metal parts in the head area
* Cardiac pacemakers
* Infusion pumps
* Heart diseases
* Increased intracranial pressure
* Pregnancy
* Cochlear implants
* Tattoos (done before the year 2000)
* Piercings (if not completely removable)
* Permanent make-up
* Nicotine or pain patches
* other MRI contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Subjective anxiety symptoms | change from T1 (baseline /study start) to T4 (immediately after treatment)
  Acrophobia Questionnaire (Cohen, 1977) with two subscales: 1) degree of anxiety (ACRO) and 2) degree of avoidance (AVOI) in height-related situations.

SECONDARY OUTCOMES:
Subjective anxiety in behavioral approach tests (BAT) | change from T1 (baseline /study start) to T4 (immediately after treatment)
  anxiety measurement by a behavioral approach test (BAT) in virtual reality (glass elevator on the outside of an high-rise building, height up to 150m) and in real life (open stairwell height up to 11,6m).
Subjective anxiety symptoms (Follow-Up) | change from T1 (baseline/ study start) to T28 (6 months follow-up)
  Acrophobia Questionnaire (Cohen, 1977) with two subscales: 1) degree of anxiety (ACRO) and 2) degree of avoidance (AVOI) in height-related situations.
Subjective anxiety in behavioral approach tests (BAT) (Follow-Up) | change from T1 (baseline /study start) to T28 (6 months follow-up)
  anxiety measurement by a behavioral approach test (BAT) in virtual reality (glass elevator on the outside of an high-rise building, height up to 150m) and in real life (open stairwell height up to 11,6m).

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Herrmann, PhD, Principal Investigator — University of Würzburg
Locations (1):
- Martin J. Herrmann, Würzburg, Germany